CLINICAL TRIAL: NCT02284633
Title: Use of a New Blood Test to Identify Response to Targeted Treatment in Patients With EGFR Mutated Lung Cancer. Evaluation in a Multicenter Study
Brief Title: Blood Sample Monitoring of Patients With EGFR Mutated Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other); Herning Hospital (Other); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Eva Boysen Hansen, MD, Aarhus University Hospital
Other Study IDs: 1-10-72-83-14; 1-16-02-431-14 (Other: Datatilsynet)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Lung Neoplasms
Keywords: EGFR mutation; Liquid biopsies; Lung cancer; erlotinib
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liquid biopsies: Bloodsamples investigating circulating tumor DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In non-small celled lung cancer (NSCLC) 10-15% of the patients harbor a mutation in the tumor's epidermal growth factor receptor (EGFR M+). This receptor is the target for treatment with erlotinib. Identification of EGFR M+ is done on a biopsy, which can be difficult to retrieve. A new blood based test identifies EGFR M+ in plasma, which makes it possible to monitor the level of EGFR M+ in the patient's blood during treatment. This enables both a closer monitoring of the treatment with erlotinib and a closer study of the resistance mechanisms that almost inevitably develop during treatment. A pilot study demonstrated that the quantity of EGFR M+ in plasma correlates to the response to treatment and might be used to predict disease progression.

Patients with EGFR M+ NSCLC referred to a participating oncology department may be enrolled in the project. The investigators expect to include 250 patients over a four-year period. Patients will receive standard treatment and follow up. Standard 1st line treatment for patients with metastatic disease is tyrosine kinase inhibitors (TKI) eg. erlotinib. A biopsy and blood sample will be retrieved before treatment with is initiated. The patient will be monitored prospectively with blood samples every 3rd-6th week both during erlotinib treatment, subsequent lines of treatment and treatment intermissions. The blood samples are analyzed for subtypes of EGFR M+ both sensitizing mutations and mutations known to drive resistance to erlotinib treatment. In the event of occurring resistance mutations or unexpected increase in quantity of sensitizing mutations clinical action will be taken; initially in the form of additional scans searching for signs of disease progression. Clinical data will be retrieved from the patient's medical journal. Patients are followed until death or at least 24 months after inclusion. Any excess biological material will be stored for up to 15 years in a bio bank for future research purposes.

We expect our results to validate the use of EGFR M+ detection and quantification via blood samples in a clinically relevant setting. The investigators expect earlier identification of disease progression to allow more cases of local treatment thus - hopefully - increasing the progression free survival. Continued blood monitoring in subsequent lines of treatment and treatment intermissions will add to our knowledge of the nature of EGFR M+ NSCLC. The sampling of biological material allows us to further investigate the biology of resistance.

DETAILED DESCRIPTION:
Background Non-small celled lung cancer (NSCLC) is one of the most common cancers in the world, and Denmark has one of the highest incidences of approximately 3800 new patients each year who are diagnosed with NSCLC, and the overall prognosis is very poor.

The EGF (epidermal growth factor) system with its known receptors and related proteins are known to play an active role in the development of cancer. In non-small cell lung cancer (NSCLC) especially EGFR has been studied. Inhibition of EGFR is associated with prolonged survival especially in patients with mutations in the EGFR (EGFR M+) 10-15% of the patients with NSCLC harbor a mutation in the tumor's EGFR. This receptor is the target for treatment with the tyrosine kinase inhibitor (TKI) erlotinib. The response rate for erlotinib treatment in EGFR M+ NSCLC is around 75% as opposed to response rates around 30% for treatment with traditional chemotherapy.

Recently, resistance mechanisms that cause progression on TKI treatment has been elucidated. The most common is the T790M mutation in EGFR, but other mechanisms such as increased MET and HER3 expression is also described. It is estimated that T790M mutations in EGFR accounts for 50% of the cases with TKI resistance development. With the exception of HER3 and MET, which is estimated to represent less than 5% of the cases with the development of resistance, are the mutations which cause the remaining 50% of cases, resistance remains unknown. The revelation of further resistance mutations hampered by the problems of obtaining biopsies when progression occurs.

Identification of EGFR M+ is done on a tumor biopsy, which can be difficult to retrieve. Furthermore a biopsy only provides information about a certain part of the one tumor site, that is tested. The investigators know that tumors especially in NSCLC is a very heterogenous group. A blood test provides us with e more overall information about the tumor mass of each specific patient. However tumor DNA is also present in blood of cancer patients in the form of circulating free DNA. A new blood based test identifies EGFR M+ in plasma, which makes it possible to monitor the level of EGFR M+ in the patient's blood during treatment. This enables both a closer monitoring of the treatment with erlotinib and a closer study of the resistance mechanisms that almost inevitably develop during treatment.

A pilot study with 23 EGFR M+ NSCLC patients demonstrated that the quantity of EGFR M+ in plasma correlates to the response to treatment and might be used to predict disease progression. In this study resistance mutations were detected between 20-300 days prior to clinical evidence of disease progression via CT scans.

Retrospective studies suggest that local treatment of oligoprogressive disease markedly increases progression free survival thus prolonging the time until a change to subsequent lines of systemic treatment is necessary.

Methods Patients with EGFR M+ NSCLC referred to one of the participating oncology departments may be offered enrollment in the project. A multicenter collaboration allows us to identify 250 EGFR M+ patients in a two-year period (200 patients with metastatic disease and 50 patients with localized disease). The EGFR mutation must be diagnosed via a diagnostic tissue sample. Patients must be over 18 years and give a written consent before entering the study. Patients can at any time withdraw their consent.

The patients will receive standard treatment and follow up. Standard 1st line treatment for patients with disseminated EGFR M+ disease is erlotinib. Standard follow up during this treatment is blood testing and clinical evaluation every 6th week and a CT scan evaluated by the RECIST criteria every 12th week. Additional tests are ordered on clinical indication. A biopsy and blood sample will be retrieved before treatment with is initiated. The patient will be monitored prospectively with blood samples (2x10 ml EDTA tubes) every 3rd-6th week both during erlotinib treatment, subsequent lines of treatment and treatment intermissions. The blood samples will be transported to the Department of Clinical Biochemistry, Aarhus University Hospital where it will be analyzed for subtypes of EGFR M+ both sensitizing mutations and mutations known to drive resistance to erlotinib treatment. Analyses are performed using the COBAS 4800 light cycler. In the event of occurring resistance mutations or unexpected increase in quantity of sensitizing mutations clinical action will be taken; initially in the form of additional scans searching for signs of disease progression. Clinical data will be retrieved from the patient's medical journal. These data include TNM status, histology, treatment modality and patient characteristics (gender, age, smoking status and performance status) Patients are followed until death or at least 24 months after inclusion.

Tissue samples will be examined retrospectively using exom sequencing. Any excess biological material will with the patients' consent be stored for up to 15 years in a bio bank at -80 degrees celsius. This allows optimal use of the material, because it will make it possible to conduct future research in the cancer field.

Aims and perspectives The overall purpose of this study is to increase our knowledge concerning molecular mechanisms - especially the development of resistance - in EGFR M+ NSCLC. Increased molecular knowledge is crucial in the development towards a more personalized cancer care. It provides us with better methods in selecting which treatment is the optimal choice for each individual patient. The investigators expect our results to validate the use of EGFR M+ detection and quantification via blood samples in a clinically relevant setting complementing CT scans in treatment evaluation. The investigators expect to be able to identify disease progression earlier than it would be possible using CT scans alone and thereby discovering more cases of oligoprogressive disease eligible for local treatment thus - hopefully - increasing the progression free survival.

The continuation of blood monitoring in subsequent lines of treatment and treatment intermissions will add to our knowledge of the nature of EGFR M+ NSCLC.

Additionally the sampling of biological material makes it possible for us to further investigate the biology of resistance.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer with a biopsy verified EGFR mutation eligible for treatment with erlotinib

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EGFR mutated lung cancer
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hansen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, DK, Denmark

IPD SHARING:
Plan to Share IPD: No